CLINICAL TRIAL: NCT05828524
Title: Outcome of Balloon Pulmonary Valvuloplasty in Patients With Congenital Pulmonary Stenosis in Terms of Reverse Right Ventricular Remodeling and Functional Exercise Capacity
Brief Title: Outcome of Balloon Pulmonary Valvuloplasty in Patients With Congenital Pulmonary Stenosis in Terms of Reverse Right Ventricular Remodelling and Functional Exercise Capacity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salah Eldin Mohammed Mostafa, Dr, Assiut University
Other Study IDs: BPVP
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease; Pulmonary Valve Stenoses
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective of 30 patients with symptomatic severe congenital valvular pulmonary stenosis who are indicated for percutaneous balloon pulmonary valvuloplasty . the aim is to

1. - evaluate electrical and mechanical remodeling of RV 6 months following balloon dilation
2. - evaluate Functional capacity using 6MWT and SaO2 before and 6 months following BPV

DETAILED DESCRIPTION:
Valvular pulmonary stenosis (PS), defined as an obstruction of blood flow at the level of the pulmonary valve, is a form of congenital heart disease, described in 0.6-0.8 out of 1000 live births.

The main physiologic effect of valvular pulmonary stenosis (PS) is an increase in Right ventricular pressure proportional to the severity of obstruction. This elevation of RV pressure is accompanied by an increase in muscle mass where hyperplasia of the muscle cells with a concomitant increase in the number of capillaries occurs. In contrast, the adult myocardium responds with hypertrophy of the existing fibers, with no change in the capillary network. Percutaneous balloon pulmonary valvuloplasty (PBPV) is the procedure of choice for uncomplicated severe or symptomatic pulmonary stenosis. the aim is to

1. - evaluate electrical and mechanical remodeling of RV 6 months following balloon dilation
2. - evaluate Functional capacity using 6MWT and SaO2 before and 6 months following BPV

ELIGIBILITY:
Inclusion Criteria:

* 1-Adult population with an age more than or equal to 16 years of age at time of procedure 2-Severe valvular Pulmonary stenosis defined as a PG max more than or equal to 64 mmHg measured by 2d echo before Procedure

Exclusion Criteria:

1. Patients with isolated supra-valvular and sub valvular pulmonary stenosis
2. Patients with peripheral pulmonary stenosis.
3. Patients with pulmonary stenosis if part of another congenital heart disease .
4. Patients with organically diseased Tricuspid valve
5. Patients with any significant shunt lesion which result in dilation in RV such as atrial septal defect.
6. Patients with right ventricular dysfunction due to arrhythmogenic right ventricular dysplasia (ARVD) or non compaction

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult population with an age more than or equal to 16 years of age at time of procedure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
reverse Right ventricular remodeling | one year
  reverse right ventricular remodeling detected by cardiac MRI and 2D echocardiography after
functional exercise capacity | one year
  assessment of functional exercise capacity by performing six minutes walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gozar L, Iancu M, Gozar H, Sglimbea A, Cerghit Paler A, Gabor-Miklosi D, Toganel R, Fagarasan A, Iurian DR, Toma D. Assessment of Biventricular Myocardial Function with 2-Dimensional Strain and Conventional Echocardiographic Parameters: A Comparative Analysis in Healthy Infants and Patients with Severe and Critical Pulmonary Stenosis. J Pers Med. 2022 Jan 6;12(1):57. doi: 10.3390/jpm12010057. PMID 35055372
- [Background] Mansour A, Elfiky AA, Mohamed AS, Ezzeldin DA. Mechanism of the right ventricular reverse remodeling after balloon pulmonary valvuloplasty in patients with congenital pulmonary stenosis: A three-dimensional echocardiographic study. Ann Pediatr Cardiol. 2020 Apr-Jun;13(2):123-129. doi: 10.4103/apc.APC_93_18. Epub 2020 Mar 20. PMID 32641883
- [Background] Deng RD, Zhang FW, Zhao GZ, Wen B, Wang SZ, Ou-Yang WB, Liu Y, Xie YQ, Pan XB. A novel double-balloon catheter for percutaneous balloon pulmonary valvuloplasty under echocardiographic guidance only. J Cardiol. 2020 Sep;76(3):236-243. doi: 10.1016/j.jjcc.2020.03.014. Epub 2020 May 22. PMID 32451153
- [Background] Behjati-Ardakani M, Forouzannia SK, Abdollahi MH, Sarebanhassanabadi M. Immediate, short, intermediate and long-term results of balloon valvuloplasty in congenital pulmonary valve stenosis. Acta Med Iran. 2013 May 30;51(5):324-8. PMID 23737317
- [Background] Alyan O, Ozdemir O, Kacmaz F, Topaloglu S, Ozbakir C, Gozu A, Korkmaz S, Toprak N. Sympathetic overactivity in patients with pulmonary stenosis and improvement after percutaneous balloon valvuloplasty. Ann Noninvasive Electrocardiol. 2008 Jul;13(3):257-65. doi: 10.1111/j.1542-474X.2008.00229.x. PMID 18713326